CLINICAL TRIAL: NCT02912377
Title: Multiple-doses, Randomised, Double-blind, Three-periods, Two-sequences Crossover Study to Assess the Immunogenicity and Pharmacodynamic Comparability of a Biosimilar Pegfilgrastim (B12019) and the Reference Product Neulasta® in Healthy Subjects
Brief Title: Immunogenicity and Pharmacodynamic of B12019 and Neulasta® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinfa Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B12019-102
Record Dates: First submitted 2016-09-19; First posted 2016-09-23 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1; B12019 / Neulasta (Experimental): 2 single doses of B12019 followed by one dose of Neulasta
  Interventions: Biological: Neulasta, B12019
- Arm 2; Neulasta / B12019 (Experimental): 2 single doses of Neulasta followed by one dose B12019
  Interventions: Biological: Neulasta, B12019

INTERVENTIONS:
Biological: Neulasta, B12019 — GCSF, Growth Colony Stimulating Factor

SUMMARY:
Multiple-doses, randomised, double-blind, three-periods, two-sequences crossover study to assess the immunogenicity and pharmacodynamic comparability of a biosimilar pegfilgrastim (B12019) and the reference product Neulasta® in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, between 18 and 55 years of age (inclusive).
2. BMI between 20.0 and 30.0 kg/m² (inclusive).
3. Weight between 60 and 100 kg (inclusive).
4. Non-smoker for at least 3 months or mild smokers with a consumption of less than 5 cigarettes (or equivalent) per day prior to study start.
5. Healthy subjects as determined by medical history, physical examination including vital signs, ECG and clinical laboratory testing.
6. Able to comply with protocol requirements, including overnight stays, blood sample collections as defined in the protocol and to participate in the entire trial period.
7. Subjects who are able and willing to give written informed consent.
8. Male subject and his female spouse/partner who is of childbearing potential must be using effective contraception starting at screening and continue throughout the clinical study period.
9. Male subject must not donate sperm starting at screening and throughout the clinical study period and for 3 months after final study drug administration.

Exclusion Criteria:

History of:

1. Evidence in the subject's medical history or in the medical examination of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, haematological, central nervous system diseases or other significant acute or chronic diseases, especially hereditary fructose intolerance, which might influence either the safety of the subject or the absorption, metabolism or excretion of the active agent under investigation.
2. Subjects with clinically relevant neurologic or psychiatric illness.
3. Subjects with clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing).
4. Previous exposure to pegfilgrastim.
5. Known hypersensitivity to Escherichia coli-derived proteins, pegfilgrastim, filgrastim or any other component of B12019 or Neulasta® as listed in section 7.2.
6. History of allergy to any recombinant protein.
7. History of cancer.
8. History of haematological disease, including sickle cell disorder.
9. History of pulmonary infiltrates or pneumonia within 6 months before the first study drug administration.
10. Known anti-drug antibodies to filgrastim or pegfilgrastim, including known antibodies to PEG as a consequence of exposure to PEG other than pegfilgrastim (e.g. cosmetics, etc.).
11. Subjects not willing or able to comply with the food and beverage restrictions (grapefruit/pomelo, starfruit, poppy seeds).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-09; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Incidence of anti-drug antibodies (ADAs) | 6 weeks
  Incidence of anti-drug antibodies over time (ADAs)
Absolute Neutrophil count (ANC) | 6 weeks
  AUEC0-last of ANC

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lissy, MD, Principal Investigator — Nuvisan GmbH, 89231 Neu-Ulm
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany